CLINICAL TRIAL: NCT00258375
Title: A Phase II Study of a Second Generation Clusterin Antisense Oligonucleotide (OGX-011) in Combination With Docetaxel in Advanced Breast Cancer
Brief Title: OGX-011 and Docetaxel in Treating Women With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I164; CAN-NCIC-IND164 (Other: PDQ); ONCOGENEX-OGX-011-06 (Other: Oncogenex Technologies); CDR0000450847 (Other: PDQ)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: custirsen sodium
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. OGX-011 may help docetaxel kill more tumor cells by making tumor cells more sensitive to the drug.

PURPOSE: This phase II trial is studying how well giving OGX-011 together with docetaxel works in treating women with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of OGX-011 and docetaxel, in terms of objective tumor response rate, in women with locally advanced or metastatic breast cancer.

Secondary

* Determine the tolerability and toxicity of this regimen in these patients.
* Determine the time to progression and overall survival of patients treated with this regimen.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive OGX-011 IV over 2 hours on days -7, -5, -3, 1, 8, and 15 of course 1 and on days 1, 8, and 15 of all subsequent courses. Patients also receive docetaxel IV over 1 hour on days 1 and 8 of all courses. Treatment repeats every 21 days* for up to 10 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Course 1 is 28 days in length and all subsequent courses (courses 2-10) are 21 days in length.

After completion of study treatment, patients are followed at 4 weeks and then periodically until disease progression.

PROJECTED ACCRUAL: Approximately 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic or locally advanced disease
  * Not curable with standard therapy
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Lesion must be outside of the previously irradiated field

    * If the sole site of disease is in a previously irradiated field, there must be evidence of disease progression or new lesions in the irradiated field
* No known CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* Absolute granulocyte count ≥ 1,500/mm^3
* PTT, PT, and INR normal
* No known bleeding disorder

Hepatic

* Bilirubin normal
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No significant cardiac dysfunction

Immunologic

* No active uncontrolled infection
* No history of serious allergic reaction to taxanes, including paclitaxel or docetaxel

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No preexisting neuropathy ≥ grade 2
* No other malignancies within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No other serious medical condition or illness that would preclude study participation
* No significant neurological disorder that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior trastuzumab (Herceptin^®) allowed

Chemotherapy

* Recovered from prior chemotherapy
* At least 6 months since prior adjuvant chemotherapy (taxanes allowed)
* At least 4 weeks since prior chemotherapy for advanced disease

  * No prior taxanes for advanced disease
* No more than 1 prior chemotherapy regimen for advanced disease
* No other concurrent chemotherapy

Endocrine therapy

* At least 1 week since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

  * Low-dose, nonmyelosuppressive radiotherapy allowed within 4 weeks before study entry at the discretion of the investigator
* No prior radiotherapy ≥ 30% of functioning bone marrow
* No concurrent radiotherapy

Surgery

* At least 3 weeks since prior major surgery and recovered (wound healing must have occurred)

Other

* More than 4 weeks since prior investigational agents or new anticancer therapy
* No concurrent therapeutic anticoagulation therapy except low-dose oral anticoagulant therapy (i.e., 1 mg of oral warfarin once a day) or low molecular weight heparin
* No other concurrent investigational therapy
* No other concurrent cytotoxic therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10-21 (Actual); Primary Completion 2007-02-23 (Actual); Study Completion 2008-09-22 (Actual)

PRIMARY OUTCOMES:
Objective response measured by RECIST criteria after accrual of 14 evaluable patients

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chia, MD, Study Chair — British Columbia Cancer Agency
Locations (5):
- Canada (5):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chia S, Dent S, Ellard SL, et al.: A phase II trial of a second generation antisense oligonucleotide (ASO) to clusterin (OGX-011) in combination with docetaxel in metastatic breast cancer (MBC): NCIC-CTG IND 164 trial. [Abstract] American Association for Cancer Research: 98th Annual Meeting, April 14-18, 2007, Los Angeles, CA. A-3512, 2007.